CLINICAL TRIAL: NCT02122133
Title: CARE: A Multicenter Case Study to Assess Radiation Exposure in Patients Treated With the Penumbra Coil 400
Brief Title: CARE: A Prospective Multicenter Case Study to Assess Radiation Exposure in Patients Treated With the Penumbra Coil 400
Acronym: CARE
Status: Terminated | Type: Observational
Why Stopped: Business decision to focus on other studies. No safety concern.
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP 7495
Record Dates: First submitted 2014-04-21; First posted 2014-04-24 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Intracranial Aneurysms
Keywords: IC aneurysms, coil embolization, PC 400, radiation exposure,
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PC 400: Patients treated with the PC 400 according to the IFU
  Interventions: Device: PC 400
- Conventional Embolic Coils: These are any approved embolic coils on the market used as part of the standard of care for treating intracranial aneurysms.
  Interventions: Device: PC 400

INTERVENTIONS:
Device: PC 400

SUMMARY:
The primary objective of this study is to gather data on the radiation exposure in patients treated with the Penumbra Coil 400™ System (PC 400) or conventional coils per their respective indications for use.This is a multicenter case review study of patients presenting with intracranial aneurysms who are treated with coil embolization therapy using the PC 400 or conventional coils. Data for each patient are collected acutely.Up to 90 patients treated with the PC 400 or conventional coils (2:1) at up to 15 centers in the USA will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in the PC 400 arm must be those treated according to the cleared indication for the PC 400 System, which includes endovascular embolization of intracranial aneurysms.
* Patients treated with conventional coils should be treated per their IFU.
* Adjunctive use of stents, balloons or liquid embolics, if considered appropriate by investigators, is allowed.

Exclusion Criteria:

* Pre-planned use of multiple coil systems and/or flow diverters.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 90 patients treated with the PC 400 or conventional coils (2:1) at up to 15 centers in the USA will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2015-05; Primary Completion 2016-10-19 (Actual); Study Completion 2016-10-19 (Actual)

PRIMARY OUTCOMES:
1. Acute radiation exposure [air kerma, kerma-area product (KAP) or dose area product (DAP), and fluoroscopic time]. | At immediate post-procedure
  Radiation exposure is measured by air kerma, kerma-area product (KAP) or dose area product (DAP), and fluoroscopic time.
2. Procedural serious adverse events | Procedural serious adverse events up until 3 days or discharge, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Abhineet Chowdhary, MD, Principal Investigator — Director of Neuro-Interventional Surgery, Overlake Hospital Medical Center, Bellevue, WA 98004
Locations (1):
- Overlake Hospital Medical Center, Bellevue, Washington, United States